CLINICAL TRIAL: NCT04200924
Title: Evaluation of Postural Control in Children With Idiopathic Toe Walking
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Lecturer in Department of Physiotheray and Rehabilitation, Bezmialem Vakif University, Bezmialem Vakif University
Other Study IDs: DT-02
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Toe Walking; Gait Disorders in Children; Postural Control; Postural Stability; Balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with idiopathic toe walking: After the demographic information, developmental history and gait information were recorded with the Evaluation Form, clinical evaluation was performed; bilateral lower extremity range of motion, flexibility, leg length measurement, and muscle strength measurement and muscular endurance tests (abdominal, back and lower extremity) will be performed. For the clinical evaluation of postural control, the Modified Balance Error Scoring System (BESS) and the Biodex Balance System for computerized evaluation will be used.
  Interventions: Other: Biodex Balance System; Other: Balance Error Scoring System (BESS)
- Healthy children: After the demographic information, developmental history and gait information were recorded with the Evaluation Form, clinical evaluation was performed; bilateral lower extremity range of motion, flexibility, leg length measurement, and muscle strength measurement and muscular endurance tests (abdominal, back and lower extremity) will be performed. For the clinical evaluation of postural control, the Modified Balance Error Scoring System (BESS) and the Biodex Balance System for computerized evaluation will be used.
  Interventions: Other: Biodex Balance System; Other: Balance Error Scoring System (BESS)

INTERVENTIONS:
Other: Biodex Balance System — For the computerized evaluation of postural control, Biodex Balance System will be used.
Other: Balance Error Scoring System (BESS) — For the clinical evaluation of postural control, the Modified Balance Error Scoring System (BESS) will be used.

SUMMARY:
The aim of this study is to evaluate postural control in children with idiopathic toe walking using computerized dynamic posturography (Biodex Balance System), which is reported to be a reliable and valid instrument for detecting changes in balance and postural control in the literature.

DETAILED DESCRIPTION:
Idiopathic toe walking (ITW) is a term used to describe the condition in which children walk with a toe-toe gait pattern in the absence of any known cause. When the literature is examined, it is reported that a possible neuromechanism of idiopathic toe walking is related to postural disorder and a deterioration of sensory information coming from the proprioceptive, vestibular, visual and / or tactile systems. The most important function of the posture is to maintain the balance during the initiation and continuation of the movement. Postural control regulates maintaining the balance and keeping the center of gravity within the body's stability limits. It includes resistance to gravity forces and mechanical support during movement. Postural control is an integral part of achieving targeted action. Although there are few studies showing the possible relationship, no studies have been found to evaluate postural control by computerized posturography in these children. In this study, we aimed to evaluate postural control in children with idiopathic toe walking using computerized dynamic posturography (Biodex Balance System).

ELIGIBILITY:
Inclusion Criteria:

* Having the diagnosis of idiopathic toe walking
* No contact with the heel in the initial contact phase of the gait
* Presence of bilateral toe walking gait
* Normal neurological and orthopedic examination results
* Achievement of independent walking before 18 months
* Absence of pervasive developmental disorder or autism

Exclusion Criteria:

* A history of BoNT-A or surgery in the last 6 months
* Presence of leg length discrepancy

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 16 children with idiopathic toe walking aged 6-15 years followed by Bezmialem Vakıf University Department of Orthopedics and Traumatology.
  16 healthy volunteers aged 6-15 years will be included in the control group.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Postural control-postural stability | 1 day
  Computerized test of postural stability with Biodex Balance System
Postural control-limits of stability | 1 day
  Computerized test of limits of stability with Biodex Balance System
Postural control-sensory integration | 1 day
  Computerized test of sensory integration with Biodex Balance System
Balance Error Scorring System-BESS | 1 day
  Clinical evaluation of postural control

CONTACTS AND LOCATIONS:
Overall Officials: Hulya N Gurses, Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)